CLINICAL TRIAL: NCT06589713
Title: Phase 1, Open Label, Single Dose Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics of Enpatoran in Male and Female Participants
Brief Title: Effect of Renal Impairment on Enpatoran Pharmacokinetics
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200569_0051; 2024-513393-22-00 (Other: EU CT Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Renal Impairment
Keywords: Renal impairment; Clinical pharmacology; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group 1 (Normal Renal Function) (Experimental)
  Interventions: Drug: Enpatoran
- Group 2 (Impaired Renal Function) (Experimental)
  Interventions: Drug: Enpatoran

INTERVENTIONS:
Drug: Enpatoran — Participants will receive a single oral dose of enpataron tablets once daily.

SUMMARY:
The purpose of this study is to assess the effect of renal impairment on the pharmacokinetics of enpatoran.

ELIGIBILITY:
Inclusion Criteria:

For Control Group 1 (Normal Renal Function):

* Medical history and physical examination without any ongoing clinically relevant findings as judged by the Investigator
* No clinically relevant findings (only minor deviations) in biochemistry, hematology, coagulation, and urinalysis examinations for the age of the participant, as judged by the Investigator; absolute lymphocyte count and absolute neutrophil count must be within normal limits

For Group 2 (Impaired Renal Function):

* Medical history and physical examination without any ongoing clinically relevant findings except for the underlying disease leading to renal impairment and consequence diseases thereof
* Chronic kidney disease
* For participants under medication, stable medication for at least 1 month
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of respiratory, gastrointestinal (including bariatric or other gastric surgeries, or other conditions that may affect drug absorption), hepatic (including hepatorenal syndrome), hematological, lymphatic, cardiovascular (such as ventricular dysfunction and congestive heart failure, cardiac arrythmia), psychiatric, neurological, genitourinary, immunological, dermatological, connective tissue diseases, or disorders that may affect the safety of the participant.
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients; history of serious allergic reactions leading to hospitalization or any other hypersensitivity reaction in general, which may affect the safety of the participant and/or outcome of the study per the Investigator's discretion
* History or presence of epilepsy, neurological disorders with seizure propensity or undiagnosed loss of consciousness, severe head trauma within 6 months or severe depression within 12 months prior to Screening), or neuropsychiatric conditions
* History of serotonin syndrome
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to Screening, which might interfere with the objectives of the study or the study procedures
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Plasma Concentrations of Enpatoran | Predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, and 48 hours postdose

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 35
Number of Participants with Abnormal Vital Signs, Laboratory Variables and 12-Lead Electrocardiogram (ECG) | Baseline and up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html